CLINICAL TRIAL: NCT01895634
Title: Reperfuse Ischemic Vessels With Endovascular Recanalization Device in JAPAN (RIVER JAPAN)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson K.K. Medical Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Rev-01
Record Dates: First submitted 2013-07-01; First posted 2013-07-10 (Estimated); Results first posted 2016-02-05 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-02

CONDITIONS: Acute Ischemic Stroke
Keywords: Ischemia; Stroke; Ischemic Stroke; Thrombectomy; Brain clot; Cerebrovascular disease; Recanalization; Revascularization; Clot Retriever; Neurovascular Intervention; Interventional Neuroradiology; neurovascular clinical trial
MeSH Terms: conditions — Ischemic Stroke; Ischemia; Stroke; Cerebrovascular Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Intervention Device: Rev-01
  Interventions: Device: Rev-01

INTERVENTIONS:
Device: Rev-01 — Treatment arm patients have used Rev-01 at least once

SUMMARY:
The main objective of this study is to document that the thrombectomy catheter (Rev-01) is effective and safe when used for revascularization in subjects with acute ischemic stroke within 8 hours of symptom onset who are ineligible for treatment with IV t-PA, or in whom treatment with IV t-PA has been ineffective.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject presenting with clinical signs and symptoms consistent with a diagnosis of acute ischemic stroke
* Onset of symptom is within 8 hours prior to treatment with Rev-01
* Treatment with IV t-PA is ineligible or ineffective
* Occluded (presenting TICI score of 0 or 1) M1 or M2 of MCA, basilar or vertebral artery, or intracranial segment of ICA, confirmed by angiography that it is accessible to the Rev-01
* NIHSS score is 8-30
* Prior to new focal disabling neurologic deficit, mRS score was 0-2
* Age from 20 y.o. to 85 y.o.
* Written informed consent to participate by subject or legal representative

Key Exclusion Criteria:

* Subject presenting; ICA dissection, Angiitis, Arterial tortuosity that would prevent the device from reaching the target vessel, Arterial stenosis > 50% that would prevent the device from reaching the target vessel, Evidence of acute intracranial hemorrhage, Evidence of mass effect or intracranial tumor, Evidence of extended early ischemic changes
* Subject with more than two major artery occluded
* Known sensitivity or ineligible to radiographic agent, or metallic allergy
* Administration of dabigatran or heparin within 48 hours preceding the onset of stroke and have an elevated APTT or PTT above twice of the normal range for the laboratory at presentation
* Known bleeding diathesis of current use of oral anticoagulants (e.g., warfarin sodium) with International Normalized Ration (INR) > 3
* Platelet count < 30,000/mm3
* Glucose < 50 mg/dL
* Severe sustained hypertension (SBP > 185mmHG or DBP > 110mmHG) refractory to pharmacological management
* Life expectancy of less than 90 days
* Pregnancy or females who are lactating
* Current participation in an investigational drug or device study
* Otherwise determined by investigator to be medically unsuitable for participation

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2013-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nobuyuki Sakai, M.D., D.M.Sc, Principal Investigator — Kobe City Medical Center General Hospital
Locations (1):
- Kobe City Medical Center General Hospital, Kobe, Hyōgo, Japan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 49
Completed | 46
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.6 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 23
Region of Enrollment [Number; unit: participants]
  Japan | 49

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Have Recanalization
Description: Proportion of subjects who had recanalization, TICI 2a or better
Time Frame: immediately post procedure
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 49
participants | 36

2. Secondary Outcome: Proportion of Subject Who Have Clot Migration/Embolization
Time Frame: immediately post procedure
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 49
participants | 0

3. Secondary Outcome: Neurological Outcome: Proportion of mRS 0-2 at 90 Days Post Procedure
Description: The Modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6, running from perfect health without symptoms to death", or similar, as accurate.
Time Frame: 90 days post procedure
Population: Missing value was not be imputed (1 missing subject was because of the missing data at 90 days by subject IC withdrawal)
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 48
participants | 30

4. Secondary Outcome: Proportion of Patients With Symptomatic and Asymptomatic Intracranial Hemorrhage (ICH)
Time Frame: 24-hour post procedure
Population: Missing value was not be imputed (1 missing subject was because of the death within 24 hours)
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 48
participants | 15

5. Secondary Outcome: All Cause Mortality
Time Frame: 90 days post-procedure
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 49
participants | 2

ADVERSE EVENTS:
Time Frame: 90 days post procedure
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 16/49
Other Adverse Events (participants affected / at risk) | 47/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=49)
Intestinal ischaemia (Gastrointestinal disorders) | 1
Rectal ulcer (Gastrointestinal disorders) | 1
Sepsis (Infections and infestations) | 1
Burns third degree (Injury, poisoning and procedural complications) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain stem infarction (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 4
Haemorrhage intracranial (Nervous system disorders) | 2
Brain oedema (Nervous system disorders) | 2
Carotid artery occlusion (Nervous system disorders) | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1
Femoral artery aneurysm (Vascular disorders) | 1
Haemorrhagic infarction (Vascular disorders) | 1
Embolism (Vascular disorders) | 1
Iliac artery occlusion (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=49)
Anaemia (Blood and lymphatic system disorders) | 8
Constipation (Gastrointestinal disorders) | 22
Diarrhoea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 6
Pyrexia (General disorders) | 3
Hepatic function abnormal (Hepatobiliary disorders) | 4
Urinary tract infection (Infections and infestations) | 8
Hypokalaemia (Metabolism and nutrition disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3
Haemorrhage intracranial (Nervous system disorders) | 11
Subarachnoid haemorrhage (Nervous system disorders) | 7
Cerebral vasoconstriction (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 7
Erythema (Skin and subcutaneous tissue disorders) | 3
Intraoperative cerebral artery occlusion (Injury, poisoning and procedural complications) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No